CLINICAL TRIAL: NCT06163794
Title: New Participatory Research Strategy and Multidimensional Phenotyping Towards Personalized Preventive Nutritional Support for Elderly People
Brief Title: Multidimensional Phenotyping Towards Personalized Preventive Nutritional Support for Elderly People
Acronym: MetabotypAGE
Status: Recruiting | Type: Observational
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Other Study IDs: INRAE-UNH-2023-1
Record Dates: First submitted 2023-11-10; First posted 2023-12-11 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Non Dependant 60 to 75 Year-old Men and Women
Keywords: personalized nutrition; deep phenotyping; inter-individual variability; metabotypes; post-prandial response to food; metabolomics; physical activity and food intake behaviors; aging; citizen science
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Collection of blood, white cell, plasma, serum, saliva, urine and stool samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Nutritional postprandial test — Metabolic responses to several test meals

SUMMARY:
There is high inter-individual variability in the response to feeding, which is determined by multiple interacting factors such as age, sex, genotype, gut microbiota, eating behaviors, physical activity or even socio-demographic factors. Original studies have recently demonstrated the possibility of predicting the postprandial response to the diet of healthy individuals on the basis of in-depth phenotyping, and of offering them foods adapted to their own metabolic capacities according to their belonging to different groups of individuals defined on the basis of the similarity of their metabolic capacities. Due to different life trajectories, inter-individual variability could be amplified upon entry into the aging period, which could explain at least in part why traditional strategies for managing chronic age-related pathologies are insufficient. The investigators aim is to propose a new strategy to better understand inter-individual variability in the response to food in the elderly based on deep phenotyping.

DETAILED DESCRIPTION:
During a first phase of the project, the investigators defined all the parameters that could be measured to realize a deep phenotyping of 150 volunteers to establish "metabotypes" and have a better understanding of the variability in the response to food. These parameters include: kinetics of change in postprandial blood glucose over a period of 4 hours following home consumption of four types of test meals (composite nutritional test); and measurement of several blood parameters either in the post-absorptive state, or in the post-prandial state, either after test meals at home, or after a fat meal in the research facility: triglycerides, insulin, C-Reactive-Protein, metabolites through open metabolomics, albumin, fatty acids, cytokines, different gene expression. Through questionnaires or tests the investigators will also assess:

food habits and preferences (with a special focus on polyphenols), olfactory and taste abilities, physical activity, muscle functionality, body composition, peripheral endothelial function and microvascular stiffness, blood pressure, oral status, cognitive function, stress and depression status, intestinal function, psycho-socio-economic status. Finally, the investigators will constitute a collection of blood, white cell, plasma, serum, saliva, urine and stool samples.

ELIGIBILITY:
Inclusion Criteria:

* - Subject with grip strength (assessed with a dynamometer) ≥16kg for women and ≥26 kg for men.
* 21 ≤ BMI ≤35
* Participant living in a rural or peri-urban area or city dweller, according to the population density grid of the Territorial Observatory (categories 3, 2 or 1 respectively).
* Cognitively able to perform tests and answer questionnaires according to the judgment of the recruiting doctor and on the basis of the Mini-Mental State Examination (MMSE)
* Available to carry out the entire protocol
* Biological assessment considered by the investigator as compatible with participation in the study,
* Subject agreeing to give written consent, and registration in the national file of volunteers who lend themselves to research
* Person subject to a social security system.

Exclusion Criteria:

* - Diabetes treated
* Sub-acute pathology (flu, gastroenteritis, bacterial infection, etc.) or trauma (fracture, surgical intervention, etc.) in the 30 days preceding inclusion.
* Hepatocellular insufficiency,
* Heart failure with decompensation,
* Renal insufficiency (clearance <30 ml/min)
* Chronic anti-inflammatory treatment, long-term corticosteroid therapy > 1 month, infiltrations
* Antibiotic treatment within 30 days prior to recruitment
* Progressive pathology at the time of inclusion (cancer, etc.)
* Gastrointestinal pathology deemed incompatible with the protocol
* Eating habits incompatible with the protocol (allergies, test food intolerances/aversions, vegan diets, ketogenic diets, etc.)
* Unstabilized thyroid diseases
* Intense physical activity (activity causing shortness of breath and sweating) > 10 hours per week
* Person who is in a period of exclusion on the National File of Healthy Volunteers
* Subject presenting a psychiatric pathology or cognitive disorders making them incapable of giving informed consent.
* Subject under guardianship, curatorship, deprived of freedoms or under the protection of justice

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy men and women aged 60 to 75 years living in a rural or peri-urban area or city dweller.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Characterize the inter-individual variability of the blood glucose postprandial response | Within the first month of study realization
  Kinetics of change in postprandial blood glucose over a period of 4 hours following home consumption of four types of test meals by continuously monitoring blood glucose

SECONDARY OUTCOMES:
Questionnaires about food habits and preferences (with a special focus on polyphenols) | Within the three months of study realization
  The investigators' objective is to have a good understanding of eating habits: estimation of precise food intake over three days but also long-term eating habits, preferences for sweet foods, salty foods, fatty foods. Participants will also be questioned about their general appetite, their neophobia, their culinary habits. An effort will be made to estimate polyphenol intake through specific questions.
Test to assess taste abilities | Within the first week of study realization
  The participants will be offered drinks containing either water (n=2) or salted water (n=8), with various concentrations of salt. The objective is to determine which drinks contain salt or not. The score will vary from 0 (only bad answers) to 8 (only good answers). A score of 8 thus means that the taste abilities are good.
Test to assess olfactory abilities | Within the first week of study realization
  Six groups of 4 vials will be presented to the participants. For each group of 4, only one vial has an odor. The first step will be to find the vial that does contain an odor. Then, the participant will have to identify the odor, choosing among 4 proposed odor. The score will increase with the number of vial found and the number of correct odor identification. It will thus vary from 0 to 8. If a participant has a score of 8, it means that he could detect each time in which vial there was an odor, and could each time identify the odor. Thus a score of 8 denotes very good olfactory abilities.
Time to walk 4 meters | Within the first two months of study realization
  The time to walk 4 m will be measured.
Time to stand up 5 times from a chair | Within the first two months of study realization
  The time to stand up 5 times from a chair will be measured.
Maximum tolerated muscle power | Within the first two months of study realization
  The maximum tolerated muscle power will be measured on a cycloergometer
Maximal isometric strength | Within the first two months of study realization
  The maximal isometric strength of the quadriceps will be measured on an isometric measuring bench.
Questionnaires about usual physical activity | Within the first two months of study realization
  The objective is to assess the amount of time usually spent by the participant for physical activity and for sedentary activities, the intensity of activities, through 28 questions. This questionnaire will give a categorical score, with 3 levels of physical activity: 1) Low: no physical activity or only low intensity activities. 2) Moderate: 3 or more days of intense activity lasting at least 20 min per day, or 5 days or more of moderate intensity activity and/or walking for at least 30 minutes per day, or 5 days or more of activity combining walking, moderate or high intensity activities. 3) Intense activity at least 3 days per week or 7 days or more of activity combining walking, moderate or high intensity activities
Measurement of total body lean mass (kg) | Within the first two months of study realization
  Lean body mass will be measured by multi frequency electrical bio impedance (Bodystat QuadScan 4000). A weak electric current is delivered to the subject through electrodes, and the voltage is measured in order to calculate impedance (resistance and reactance) of the body. Most body water is stored in muscle. Therefore, if a person is more muscular there is a high chance that the person will also have more body water, which leads to lower impedance. Using the weight of the participant, through calibration curves, the system then calculates total body water, total body fat mass, and total body lean mass.
Measurement of total body fat mass (kg) | Within the first two months of study realization
  Fat body mass will be measured by multi frequency electrical bio impedance (Bodystat QuadScan 4000). A weak electric current is delivered to the subject through electrodes, and the voltage is measured in order to calculate impedance (resistance and reactance) of the body. Most body water is stored in muscle. Therefore, if a person is more muscular there is a high chance that the person will also have more body water, which leads to lower impedance. Using the weight of the participant, through calibration curves, the system then calculates total body water, total body fat mass, and total body lean mass.
Measurement of peripheral endothelial function (RHI, %) | Within the first week of study realization
  Peripheral endothelial function of the participants will be assessed by tonometry using the Endo-PAT X system (Itamar Medical Ltd) before and after induction of post-occlusive reactive hyperemia. Endothelium-induced changes in vascular tone are measured at the fingertip using a pair of single-use plethysmographic sensors. The result obtained is the Reactive Hyperemia Index (RHI, %) which corresponds to the ratio between the amplitudes of the PAT® (Peripheral Arterial Tonometry) signal during hyperemia and the basal amplitudes of the occluded side, normalized by the values of the control arm. The values will be considered as normal if inferior to 1.67, and abnormal if higher than 1.67.
Measurement of microvascular stiffness (Augmentation Index) | Within the first week of study realization
  Microvascular stiffness (=Augmentation Index) of the participants will be assessed by tonometry using the Endo-PAT X system (Itamar Medical Ltd). Augmentation Index (AI) will be calculated from the shape of the pulse wave recorded in basal conditions. This measurement is a recognized marker of cardiovascular risk. The AI value is inversely proportional to the stiffness of the vessels. The scale of the measurement is the following:
  Values between 20-80: healthy degree of arterial flexibility. Values between 81-100 : increased cardiovascular risk Values over 100: high cardiovascular risk.
Assessment of oral status | Within the first two months of study realization.
  Oral status will be assessed through the Nordic Orofacial Test - Screening (NOT-S), which is a screening and evaluation tool for orofacial motor dysfunctions and disorders. It includes two parts: 1) "Maintenance" part containing 6 sections: sensory function, breathing, habits, chewing and swallowing, drooling, and dry mouth (I-VI); 2) "Examination" part comprising 6 sections: face at rest, nasal breathing, facial expression, function of the masticatory muscles and jaws, oral motor functions, and articulation of speech. The NOT-S total score ranges from 0 (no dysfunction) to 12 (high dysfunction). For each section, from the moment the subject answers "Yes" to one of the questions, the box is checked and results in a score of 1 in the last right column of the questionnaire.
Assessment of cognitive function | Within the first week of study realization
  The cognitive abilities of the participants will be assessed using the CANTAB®, using a computer under supervision. This method makes it possible to assess 1) episodic memory; 2) verbal recognition memory, that is, immediate and delayed memory for verbal information; 3) Spatial working memory, which requires the retention and manipulation of visuospatial information. 4) The spatial span task (CANTAB spatial spam), which evaluates the maximum amount of information that the subject is capable of recalling after a single presentation.
Assessment of depression status | Within the first week of study realization.
  Participants' depressive nature will be assessed using the Geriatric Depression Scale (GDS) test. It is a self-questionnaire which contains 15 items, each with a binary Yes-No response. It is a commonly used tool to assess the presence of depressive symptoms in older adults. A score of 0 to 5 is considered normal. A score between 5 and 9 indicates a high likelihood of depression, and a score between 10 and 15 almost always indicates depression.
Assessment of socio-economic status | Within the three months of study realization
  The socio-economic status of participants will be assessed using the EPICES scale (Évaluation de la Précarité et des Inégalités de santé dans les Centres d'Examens de Santé) which was developed in France by the National Institute of Prevention and Education for Health . This scale is used in public health to assess the social precariousness of individuals, which takes into account the multidimensional nature of precariousness. The main interest of the EPICES score consists of understanding populations which, while escaping the traditional administrative indicators of precariousness, present the same health risks. The EPICES score is based on 11 questions which summarize 90% of a subject's precarious situation. The answer to each question is assigned a coefficient, the sum of the 11 answers gives the EPICES score. The score is continuous, it varies from 0 (absence of precariousness) to 100 (maximum of precariousness).
Assessment of self-esteem | Within the three months of study realization
  Participants' self-esteem will be assessed using the Rosenberg Self-Esteem Scale. It is a psychometric tool widely used in psychology research, social sciences and clinical settings. It consists of 10 questions to which respondents are asked to indicate their degree of agreement or disagreement using a 4-point Likert scale, ranging from "strongly disagree" to "strongly agree". The questions are designed to assess overall self-perception and personal esteem. The score between 10 and 40 which are interpreted according to specific thresholds.Higher scores indicate higher self-esteem.
Assessment of intestinal function | Within the first month of study realization
  To have a better understanding of the characteristics of the participants' intestinal function, they will have to complete an intestinal transit diary. Such a diary is a tool used to record a person's stool habits and characteristics over a period of time. It is often used in the field of gastroenterology and nutrition to assess the functioning of the digestive system. Participants will note every day for 15 days: the frequency of stools, noting each time the time they had a bowel movement, as well as the consistency of stools based on the Bristol visual scale. which categorizes 7 types of stools, ranging from the hardest to the softest. Experts consider types 1 and 2 to be uncharacteristically hard and indicative of constipation, while types 6 and 7 are unusually loose and may indicate diarrhea. Medical professionals generally consider types 3, 4, and 5 to be the most typical. Overall, a qualitative assessment of intestinal function will be made, with no calculated score.
Stool collection | Within the first month of study realization
  One sample of stool will be taken and analyzed by metagenomic.
Measurement of plasma insulin levels (micro U / mL) | Within the first two months of study realization
  These measurements will be made 1) in the post-absorptive state, 2) after the ingestion of 4 standards test meals, 3) after the ingestion of a sweet and fatty meal.
Measurement of plasma triglycerides levels (mg / dL) | Within the first two months of study realization
  These measurements will be made 1) in the post-absorptive state, 2) after the ingestion of 4 standards test meals, 3) after the ingestion of a sweet and fatty meal.
Measurement of plasma C Reactive Protein (mg / L) | Within the first two months of study realization
  These measurements will be made in the post-absorptive state.
Measurement of plasma amino acid levels (µMol) | Within the first two months of study realization
  These measurements will be made 1) in the post-absorptive state 2) after the ingestion of a protein rich test meal.
Measurement of plasma metabolite through open metabolomics | Within the first two months of study realization
  These measurements will be made 1) in the post-absorptive state 2) after the ingestion of a sweet and fatty meal.
Measurement of plasma free fatty acids (mg / L) | Within the first two months of study realization
  These measurements will be made 1) in the post-absorptive state 2) after the ingestion of a sweet and fatty meal.
Measurement of plasma cytokines (U / L) | Within the first two months of study realization
  These measurements will be made 1) in the post-absorptive state 2) after the ingestion of a sweet and fatty meal.
Measurement of plasma albumin (g / L) | Within the first two months of study realization
  These measurements will be made in the post-absorptive state
Measurement of various gene expression in peripheral blood mononuclear cells isolated from blood samples. | Within the first two months of study realization
  These measurements will be made in the post-absorptive state

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle Pichering, Pr, Principal Investigator — Centre d'Investigation Clinique
Locations (3):
- France (3):
  - Pic / Cic-Inserm 1405, Clermont-Ferrand, France
  - Plateforme d'Exploration de la Mobilité (CHU Clermont-Ferrand), Clermont-Ferrand
  - Centre de Recherche en Odontologie Clinique, Faculté de Chirurgie Dentaire, Clermont-Ferrand

IPD SHARING:
Plan to Share IPD: Yes
Sharing of all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after publication, and for as long as necessary after that
Access Criteria: The data will be shared with any researcher who requests it by email following publication.

REFERENCES:
- [Background] Ordovas JM, Ferguson LR, Tai ES, Mathers JC. Personalised nutrition and health. BMJ. 2018 Jun 13;361:bmj.k2173. doi: 10.1136/bmj.k2173. PMID 29898881
- [Background] Berry SE, Valdes AM, Drew DA, Asnicar F, Mazidi M, Wolf J, Capdevila J, Hadjigeorgiou G, Davies R, Al Khatib H, Bonnett C, Ganesh S, Bakker E, Hart D, Mangino M, Merino J, Linenberg I, Wyatt P, Ordovas JM, Gardner CD, Delahanty LM, Chan AT, Segata N, Franks PW, Spector TD. Human postprandial responses to food and potential for precision nutrition. Nat Med. 2020 Jun;26(6):964-973. doi: 10.1038/s41591-020-0934-0. Epub 2020 Jun 11. PMID 32528151
- [Background] Zeevi D, Korem T, Zmora N, Israeli D, Rothschild D, Weinberger A, Ben-Yacov O, Lador D, Avnit-Sagi T, Lotan-Pompan M, Suez J, Mahdi JA, Matot E, Malka G, Kosower N, Rein M, Zilberman-Schapira G, Dohnalova L, Pevsner-Fischer M, Bikovsky R, Halpern Z, Elinav E, Segal E. Personalized Nutrition by Prediction of Glycemic Responses. Cell. 2015 Nov 19;163(5):1079-1094. doi: 10.1016/j.cell.2015.11.001. PMID 26590418
- [Background] Hillesheim E, Ryan MF, Gibney E, Roche HM, Brennan L. Optimisation of a metabotype approach to deliver targeted dietary advice. Nutr Metab (Lond). 2020 Sep 29;17:82. doi: 10.1186/s12986-020-00499-z. eCollection 2020. PMID 33005208
- [Background] Delude CM. Deep phenotyping: The details of disease. Nature. 2015 Nov 5;527(7576):S14-5. doi: 10.1038/527S14a. No abstract available. PMID 26536218
- [Background] de Toro-Martin J, Arsenault BJ, Despres JP, Vohl MC. Precision Nutrition: A Review of Personalized Nutritional Approaches for the Prevention and Management of Metabolic Syndrome. Nutrients. 2017 Aug 22;9(8):913. doi: 10.3390/nu9080913. PMID 28829397